CLINICAL TRIAL: NCT03195049
Title: Complications of Exchange Transfusion in Neonates
Acronym: COET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Zanaty, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COET
Record Dates: First submitted 2017-06-15; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Kernicterus
Keywords: hyperbilirubinemia; kernicterus
MeSH Terms: conditions — Kernicterus; Hyperbilirubinemia | interventions — Blood Grouping and Crossmatching; Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood group (Experimental): blood is collected for maternal and infant blood group,complete blood count,before, during and after the procedure of exchange transfusion .
  Interventions: Diagnostic Test: blood group,complete blood count
- serum bilirubin estimation (Experimental): estimation of serum bilirubin before, during and after the procedure of exchange transfusion .
  Interventions: Diagnostic Test: blood group,complete blood count

INTERVENTIONS:
Diagnostic Test: blood group,complete blood count — measure levels of total and direct bilirubin before, during and after the procedure of exchange transfusion
  Other Names: measure levels of total and direct bilirubin

SUMMARY:
Exchange transfusion is effective and considered to be safe procedure ; however, it is not without risks. Complications have been reported and mortality rates vary from 0.5 to 3.3%. therefore ,the current recommendation for performing exchange transfusion are based on balance between the risks of encephalopathy and complications related to the procedure .

DETAILED DESCRIPTION:
About 60% of term and 80% of preterm infants have clinical jaundice in the first week after birth but only 2% to 16% of them develop severe hyperbilirubinemia (total serum bilirubin > 25mg/dl) ,which is an emergency because it may cause neonatal bilirubin encephalopathy (kernicterus), which can result in death or irreversible brain damage in survivor.

Exchange transfusion is the standard method of therapy for immediate treatment of severe hyperbilirubinemia and prevention of kernicterus. Although the frequency of neonatal exchange transfusion has declined markedly in the past two decades, this procedure is still performed in many countries, especially in those with a high incidence of neonatal hyperbilirubinemia.

Exchange transfusion is effective and considered to be safe procedure ; however, it is not without risks. Complications have been reported and mortality rates vary from 0.5 to 3.3%. therefore,the current recommendation for performing exchange transfusion are based on balance between the risks of encephalopathy and complications related to the procedure .

Most of these complications are transient, such as severe thrombocytopenia, apnea, hypocalcemia , bradycardia, and hyperkalemia and recovery is expected along with appropriate care and follow up. But serious complications and even death can occurs due to cardiovascular collapse during exchange , necrotizing enterocolitis, bacterial sepsis, and pulmonary hemorrhage that can be avoided by careful cardio-pulmonary and oxygen saturation monitoring.

ELIGIBILITY:
Inclusion Criteria:

* All preterm and full term neonates who need exchange transfusion

Exclusion Criteria:

* Neonatal sepsis
* Congenital anomalies

Ages: 1 Day to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
serum bilirubin estimation | 2 days
  estimation of serum bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Ab Mohamed, Professor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steiner LA, Bizzarro MJ, Ehrenkranz RA, Gallagher PG. A decline in the frequency of neonatal exchange transfusions and its effect on exchange-related morbidity and mortality. Pediatrics. 2007 Jul;120(1):27-32. doi: 10.1542/peds.2006-2910. PMID 17606558
- [Result] Bhutani VK, Johnson LH, Keren R. Diagnosis and management of hyperbilirubinemia in the term neonate: for a safer first week. Pediatr Clin North Am. 2004 Aug;51(4):843-61, vii. doi: 10.1016/j.pcl.2004.03.011. PMID 15275978